CLINICAL TRIAL: NCT00936299
Title: Bupropion for ADHD in Adolescents With Substance Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0178; R01DA022284 (NIH)
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Nicotine Dependence; Cannabis Use Disorder
Keywords: Adolescents; Substance Use Disorder; Attention Deficit Hyperactivity Disorder; Cognitive Behavioral Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Tobacco Use Disorder; Substance-Related Disorders | interventions — Bupropion; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion + cognitive behavioral therapy (Active Comparator): Adolescents with ADHD, nicotine dependence, and cannabis use disorders receive bupropion + CBT.
  Interventions: Drug: Bupropion
- Placebo + cognitive behavioral therapy (Placebo Comparator): Adolescents with ADHD, nicotine dependence, and cannabis use disorders receive placebo + CBT.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion — Bupropion (target dose 300 mg/day) + cognitive behavioral therapy; matched placebo + cognitive behavioral therapy
  Arms: Bupropion + cognitive behavioral therapy
Other: Placebo
  Other Names: Sugar Pill
  Arms: Placebo + cognitive behavioral therapy

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is one of the most common co-occurring psychiatric disorders (30-50%) in adolescents with substance use disorders (SUD). Yet, little is known about the safety and efficacy of medications for ADHD in adolescents with SUD, since such youths have been excluded from most medication trials. Clinicians are therefore understandably reluctant to treat ADHD in substance abusing adolescents, often first referring such youths to substance treatment. Untreated ADHD is associated with poorer substance treatment outcomes. We address this research gap by proposing a randomized controlled trial of bupropion vs placebo in 130 adolescents (13-19 years) with Diagnostic and Statistical Manual (DSM IV) ADHD, nicotine dependence and cannabis use disorder (not excluding other SUD). Participants in both bupropion and placebo treatment groups will receive weekly individual manualized-standardized cognitive behavioral therapy (CBT) targeting SUD (at no cost to them) throughout the 16 weeks of the medication trial. Bupropion also is effective in treating nicotine dependence in adults; the majority of adolescents with marijuana and other drug abuse also smoke tobacco. More recent research in adults indicates that bupropion may reduce craving and use of other substances of abuse (e.g. methamphetamine, cocaine). It's possible impact on cannabis use disorder (the addiction for which most teens are referred to treatment) has not yet been evaluated. However since all drugs of abuse have a final common pathway leading to addiction via action in the so called brain reward system (ventral tegmental area (VTA), accumbens) -an important secondary aim is to evaluate bupropion's potential impact on craving and use of marijuana (MJ) in addition to its known similar action on nicotine.

DETAILED DESCRIPTION:
Research has shown that bupropion is a safe and effective treatment for both ADHD and nicotine dependence in individuals without SUD, and newer research provides empirical support for its unique pharmacotherapeutic properties and potential for treating other addictive disorders (e.g., methamphetamine dependence, pathological gambling). No controlled studies have yet evaluated bupropion's safety and efficacy for ADHD and SUD (including nicotine and cannabis) in adolescents. The lack of research on the safety and efficacy of medications in adolescents with SUD and psychiatric comorbidities contributes to a serious lack of integrated treatment for commonly co-occurring mental health and substance problems in community-based adolescent drug treatment programs. This then contributes to poorer treatment outcomes and prognosis for the large number of comorbid youths with substance abuse and mental health problems that significantly impact public health. The specific aims of the proposed study will address this research gap by conducting a 16-week randomized controlled trial of bupropion vs. placebo to evaluate the safety and efficacy of this low abuse potential medication on ADHD, nicotine dependence, and cannabis use disorders (not excluding other SUD) in 130 adolescents (13-19) receiving concurrent outpatient substance treatment (CBT). The study design and analytic approach will enable assessment of the complex inter-relationship between change in ADHD, depression/dysphoria (and other psychiatric symptoms) and change in nicotine, cannabis and other substance use within and between treatment groups. Thus, the study addresses important research gaps in at least two priority areas of the National Institute on Drug Abuse/ National Institutes of Health(NIDA/NIH) research agenda: 1) research on effective treatments for adolescents with addiction and psychiatric comorbidity, and 2) medications development research for nicotine and cannabis use disorders in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 13 and 19, with a parent or legal guardian available to complete parental assessments for minors;
* Meet DSM-IV diagnostic criteria for ADHD on the K-SADS-PL;
* Schedule for Affective Disorders and Schizophrenia score ≥ 22 on the DSM-IV ADHD symptom checklist;
* Meet DSM-IV criteria for nicotine dependence (and/or cut off score of >3 on modified Fagerstrom);
* Meet DSM-IV criteria for cannabis abuse or dependence on the Kiddie-Sads-Present and Lifetime (K-SADS-PL);
* Have used marijuana at least 5 of the past 30 days;
* Have used nicotine at least 15 days out of the past 30 days;
* Be medically healthy;
* If female, subjects must use an effective birth control method if sexually active.

Exclusion Criteria:

* Current or past psychosis;
* Bipolar I or II disorder;
* A first-degree relative with bipolar I disorder;
* A lifetime history of seizure disorder;
* Any other chronic or serious medical illnesses;
* A lifetime history of eating disorder;
* Current pregnancy;
* Previous clinically significant adverse reaction to bupropion;
* The need to take other psychotropic medications at the time of study entry. Patients may have had previous psychotherapy or pharmacotherapy for ADHD or other co-morbidity but cannot have been on psychotropic medication for at least one month prior to study entry;
* Active participation in substance abuse treatment or mental health treatment (including outpatient, day-treatment, residential, or inpatient) within 28 days prior to signing consent;
* Non-English speaking (due to the difficulty in translating the additional materials given to the subjects);
* Cognitively impaired or of low intelligence;
* Breastfeeding;
* Current use of other psychotropic medications including nicotine replacement therapy;
* Current opiate dependence.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula D Riggs, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Adolescent Clinical Research, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupropion + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy
Started | 53 | 52
Completed | 40 | 40
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.8 (1.5) | 17.8 (1.6) | 17.8 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 46 | 46 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 5 | 12
  White | 28 | 31 | 59
  More than one race | 5 | 13 | 18
  Unknown or Not Reported | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 15 | 27
  Not Hispanic or Latino | 41 | 37 | 78
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change in ADHD Rating Scale (ADHD-RS) Total Score
Description: DSM-IV ADHD Rating Scale (ADHD-RS) Total Score (clinician administered/adolescent informant). Total scale range 0-54, higher is greater severity.
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bupropion + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy
Number analyzed (Participants) | 53 | 52
units on a scale | -14.2 [-17.1 to -11.4] | -13.8 [-16.6 to -11.1]

2. Primary Outcome: Change in Number of Days of Cigarette Smoking in Past 28 Days
Description: The number of days of cigarette smoking in the past 28 days was ascertained based on adolescent self-report using calendar-based timeline follow back procedures. Mean number of days of past 28-day cigarette smoking at baseline was compared to mean number of days of past 28-day cigarette smoking at end of 16-week trial.
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: days of use
Groups:
- Placebo + Cognitive Behavioral Therapy: Adolescents with ADHD, nicotine dependence, and cannabis use disorders receive placebo + CBT.
  Placebo
Arm/Group | Bupropion + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy
Number analyzed (Participants) | 53 | 52
days of use | -4.1 [-6.7 to -1.5] | -2.7 [-5.3 to -0.1]

3. Secondary Outcome: Change in Number of Days of Cannabis Use in Past 28 Days
Description: The number of days of cannabis use in the past 28 days was ascertained based on adolescent self-report using calendar-based timeline follow back procedures. Mean number of days of past 28-day cannabis use at baseline was compared to mean number of days of past 28-day cannabis use at end of 16-week trial.
Time Frame: Baseline, 16 Weeks
Measure: Mean (95% Confidence Interval); unit: days of use
Arm/Group | Bupropion + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy
Number analyzed (Participants) | 53 | 52
days of use | -4.7 [-7.6 to -1.8] | -6.5 [-9.4 to -3.6]

ADVERSE EVENTS:
Arm/Group | Bupropion + Cognitive Behavioral Therapy | Placebo + Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 2/53 | 2/52
Other Adverse Events (participants affected / at risk) | 45/53 | 45/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion + Cognitive Behavioral Therapy (N=53) | Placebo + Cognitive Behavioral Therapy (N=52)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) — Participant hospitalized for alleged bipolar (mania) episode.
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1) — Participant hospitalized overnight for tonsillitis.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Participant hospitalized for two days for pneumonia.
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Participant hospitalized for possible head injury due to a fight.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion + Cognitive Behavioral Therapy (N=53) | Placebo + Cognitive Behavioral Therapy (N=52)
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Anger (Psychiatric disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Decreased appetite (General disorders) | 7 | 5
Depression (Psychiatric disorders) | 9 | 10
Dizziness (Nervous system disorders) | 4 | 3
Elevated blood pressure (General disorders) | 7 | 5
Elevated pulse (General disorders) | 21 | 13
Headache (General disorders) | 12 | 14
Insomnia (General disorders) | 7 | 10
Irritability (Nervous system disorders) | 7 | 10
Low blood pressure (General disorders) | 3 | 3
Low pulse (General disorders) | 3 | 5
Migraine (General disorders) | 4 | 2
Muscle pain/soreness (Musculoskeletal and connective tissue disorders) | 10 | 9
Nausea (Gastrointestinal disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Stomache ache (Gastrointestinal disorders) | 8 | 6
Vomited (Gastrointestinal disorders) | 7 | 7
Weight gain (General disorders) | 14 | 19
Weight loss (General disorders) | 15 | 14
Worse headache (General disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Actual study enrollment N=105 was less than targeted enrollment N=130. Thus, negative results should be interpreted with caution because the study was likely underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No